CLINICAL TRIAL: NCT06806280
Title: Respiration Efter Hysterektomi Med Robotassisterad Laparoskopi- REHYR
Brief Title: Respiration After Robot Assisted Laparoscopic Hysterectomy
Acronym: REHYR
Status: Recruiting | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: FoU in VGR ID: 284148
Record Dates: First submitted 2025-01-23; First posted 2025-02-04 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-03

CONDITIONS: Cancer Uterus Cervix
Keywords: respiration; hysterctomy; robot assisted surgery
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: The study will include a consecutive series of 80 women ≥18 years of age undergoing robotic-assisted laparoscopic hysterectomy for endometrial cancer or endometrial intraepithelial neoplasia.
  Exclusion criteria are: cognitive impairment and difficulty understanding Swedish or English instructions.

SUMMARY:
The study will investigate how respiratory function is affected by robot-assisted surgery. Previous studies have investigated the impact after open and laparoscopic surgery, but there are no studies yet after robot-assisted surgery.

80 women undergoing robot-assisted hysterectomy will undergo measurements of lung function and oxygen saturation before and after the operation.

DETAILED DESCRIPTION:
It is well known that respiration is affected during surgery under general anesthesia. Despite optimal ventilation in a respirator during the procedure, lung volume decreases, leading to atelectasis. Other effects include increased secretions in the airways, while ciliary function deteriorates. After surgery performed under general anesthesia, the patient therefore often develops hypoventilation. This can largely be explained by lingering effects of anesthetics, reduced lung volumes, atelectasis, pain and immobilization.

In a previous study, lung effects have been studied in open and laparoscopic surgery, including after hysterectomy. With the development of robotic surgery and operations on patients with an increasing number of risk factors, complementary studies are needed.

The aim of the study is to investigate changes in lung function during robot-assisted laparoscopic surgery due to uterine cancer or endometrial intraepithelial neoplasia in the uterus, and to search for predictors of low lung volume, hypoxia and pneumonia.

A consecutive series of 80 patients undergoing robot-assisted hysterectomy will be included in the study.

At the preoperative visit, a dynamic spirometry (Easyone, ndd, Medical Technologies, Switzerland) is performed in a sitting position according to international guidelines. Before the test, oxygen saturation will be measured with a finger probe. In addition, patients will assess their lung function on a visual analogue scale

Postoperatively, patients will undergo the same spirometry 2-3 hours after arrival at the postoperative ward, before the first mobilization. The test will be performed while sitting in bed with the head of the bed elevated at 60˚ and with optimal pain relief (VAS<4). Pre-test pain assessment will be recorded as well as the patient's assessment of their lung function. The day after surgery, the same test will be performed again (including assessment of pain and lung function) in the morning before and after mobilization to walk in the room. During the hospitalization, mobilization and any breathing exercises are recorded on a special protocol.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age undergoing robotic-assisted laparoscopic hysterectomy for endometrial cancer or endometrial intraepitelial neoplasty..

Exclusion Criteria:

* cognitive impairment and difficulty understanding Swedish or English instructions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women develop uterus cancer
Study Population: Sahlgrenska University hospital, Gothenburg, Sweden
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity, FVC | Up to the first day after surgery
  A spirometry including FVC will be performed in the sitting position according to international guidelines.

SECONDARY OUTCOMES:
Oxygen saturation | Up to the first day after surgery
  Oxygen saturation will be performed via a finger probe.
Forced expiratory volume during one second, FEV1 | Up to the first day after surgery
  A spirometry including FEV1 will be performed in the sitting position according to international guidelines.

OTHER OUTCOMES:
Patient assessed overall lung function | Up to the first day after surgery
  The patients will assess their overall lung function on a study-specifik numeric rating scale from 0-10 (best)
Peak Expiratory Flow, PEF | Up to the first day after surgery
  A spirometry including PEF will be performed in the sitting position according to international guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided